CLINICAL TRIAL: NCT01269411
Title: Phase I Pharmacodynamic and "High Content" Study of the Gamma-Secretase Inhibitor RO4929097 in Patients With Recurrent Malignant Gliomas (MGs) Targeting p75NTR to Inhibit Brain Tumor Initiating Cells (BTICs) and Recurrent Invasive Gliomas
Brief Title: RO4929097 in Treating Patients With Recurrent Invasive Gliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02565; PHL-075; N01CM00032 (NIH); CDR0000691784 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2010-12-31; First posted 2011-01-04 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- Treatment (RO4929097 and surgery) (Experimental): PART A: Patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  PART B: Patients receive oral RO4929097 once daily on days 1-7 and undergo surgery on day 8. Beginning 28 days later, patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Other Names: R4733; RO4929097
Procedure: therapeutic conventional surgery — Undergo surgery
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative

SUMMARY:
This phase I trial is studying the side effects and best dose of RO4929097 in treating patients with recurrent invasive gliomas. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine, in patients with recurrent MGs (many of whom receive dexamethasone, a moderate CYP3A4 inducer), the safety and maximum-tolerated dose of RO4909297 administered at 2 dose levels.

II. Determine the pharmacokinetics, intratumoral drug concentration, target modulation, and evidence of any treatment effect in the malignant glioma tumor tissue by R04929097 administered at the dose found in Part A.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetic (PK) profile of RO4909297 in patients with recurrent MGs (many of whom receive dexamethasone, a moderate CYP3A4 inducer).

II. Determine the progression-free survival of patients with recurrent malignant glioma following treatment with R04929097.

III. Determine if the RPTD dose of RO4929097 significantly inhibits p75^NTR cleavage and processing.

IV. Determine the effects of RO4929097 on the establishment and growth of BTIC cultures in neurosphere growth conditions, effects on proliferation, ability to self-renewal, and ability to differentiate along lineage-specific pathways.

V. Determine the ability of RO4929097 to inhibit Notch signaling, by assessing downstream target activation, in glioma tissue of patients with recurrent MG.

VI. Determine the association between a number of serum, tumor, and BTIC markers and response to R04929097.

OUTLINE: This is a multicenter, dose-escalation (part A) study followed by an open-label (part B) study.

PART A: Patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

PART B: Patients receive oral RO4929097 once daily on days 1-7 and undergo surgery on day 8. Beginning 28 days later, patients receive oral RO4929097 once daily on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Post resection tumor specimens are collected for correlative studies, including pharmacokinetic and biomarker assays.

After completion of study therapy, patients are followed up at 30 days and then every 3 month for up to 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiographic progression of a histologically confirmed glioblastoma, high-grade astrocytoma, NOS, anaplastic mixed oligo-astrocytoma, or anaplastic oligodendroglioma

  * In patients that present radiographic evidence of progression after concurrent treatment with radiation and low-dose temozolomide, diagnosis of progression should be made after at least 2 cycles of monthly temozolomide in order to rule out pseudoprogression
  * Secondary MGs (evolving from a prior low-grade glioma) can be included as long as they are considered malignant in the latest resection
* Patients must have at least one enhancing lesion that can be accurately measured as > 1 X 1 cm on a MRI
* Prior treatment must include radiotherapy (with or without temozolomide)

  * No limit to the number of prior recurrences or surgeries
* For Part B only, surgical resection should be considered a reasonable therapeutic option for a patient that can tolerate surgical resection

  * Patients with multifocal disease can be included as long as resection is considered a reasonable option to manage the nodule that is progressing
  * There must be sufficient tissue available (minimum from a 1 X 1 cm lesion) for a biopsy to be taken during surgery
* There must be sufficient tissue available for evaluation of p75^NTR status from a prior surgery (using immunohistochemistry on fixed tissue or, in uncommon cases in which frozen tissue is available from a prior surgery, western blot) (part B)
* ECOG performance status < 2 (Karnofsky > 50%)
* Life expectancy of greater than 4 weeks
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* Hemoglobin > 90 g/L (or > 9 g/dL)
* Total bilirubin < 2.0 mg/dL
* BUN < 25 mg/dL
* AST/ALT < 3 X institutional upper limit of normal
* Creatinine within institutional normal limits OR creatinine clearance > 60 mL/min
* No major medical illnesses or psychiatric impairments that, in the investigator's opinion, would prevent administration or completion of protocol therapy
* Not pregnant or nursing
* Negative serum pregnancy test
* Fertile patients must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, during, and for 12 months after completion of study therapy
* Able to swallow pills
* Patients with a history of seizures need to have had no generalized seizures in the last month prior to entering the study
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* Patients who are serologically positive for hepatitis A, B, or C, and have a resulting positive serological test, or have a history of liver disease, other forms of hepatitis, or cirrhosis are ineligible
* No uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia, or hypokalemia (within 7 days prior to study treatment), despite adequate electrolyte supplementation
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Baseline QTc ≤ 450 msec (male) or QTc ≤ 470 msec (female)
* No history of risk factors for QT interval prolongation, including, but not limited to, family or personal history of long QT syndrome, recurrent syncope without known etiology, or sudden unexpected death
* No history of torsades de pointes or other significant cardiac arrhythmias or the need for concomitant meds with known potential to prolong QT interval or antiarrhythmics
* Use of food that may interfere with the metabolism of RO4929097 is prohibited, including grapefruit or grapefruit juice
* Patients must have recovered from the effects of any prior treatment (systemic chemotherapy/radiotherapy) or surgery (<CTCAE grade 2 toxicities related to prior therapy)
* Patients who have had chemotherapy, surgery, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study are not eligible
* Patients may not be receiving any other investigational agents
* Patients cannot be receiving enzyme-inducing anti-epileptic drugs (EIAEDs)

  * If previously treated with EIAEDs, patients must have been switched to non-EIAEDs 4 weeks prior to starting RO4929097
  * Enzyme-inducing antiepileptic drugs (EIAEDs) include: carbamazepine (Tegretol); oxcarbazepine (Trileptal); phenobarbital (or derivatives); phenytoin (Dilantin)
  * 3.1.10.2 Non enzyme-inducing Antiepileptic Drugs (Non-EIAEDs) include: clobazam (Frisium); clonazepam (Rivotril); gabapentin (Neurontin); levetiracetam (Keppra); lamotrigine (Lamictal); topiramate (Topamax)
* No concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4

  * Even though dexamethasone is a moderate inducer of CYP3A4, patients may remain on dexamethasone at the lowest dose possible
* Stable or decreasing steroid dose within 5 days prior to registration required
* No medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)
* No other investigational or commercial agents or therapies may be administered with the intent to treat the patient's malignancy
* No re-irradiation (any technique) is allowed
* If a patient elects to have a new resection of his/her tumor in the absence of progression of the disease, treatment will be discontinued and no re-challenge will be allowed after this additional surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) defined as the dose level in which less than or equal to 1 out of 6 patients experience dose limiting toxicity (DLT) assessed using NCI CTCAE version 4.0 | 21 days
Pharmacokinetic (PK) profile of RO4909297 | Pre-dose, 1, 2, 4, 8, and 24 hours

SECONDARY OUTCOMES:
Progression-free survival following treatment with R04929097 | From registration to time of progression or death, whichever occurs first, assessed up to 12 months
  The Kaplan-Meier method will be used.
Inhibition of p75NTR cleavage and processing | Up to 12 months
  Descriptive statistics, such as the mean, median and range, will be used to summarize the marker across patients. The Wilcoxon signed-rank and rank sum tests will be used.
Establishment and growth of BTIC cultures in neurosphere growth conditions, effects on proliferation, ability to self-renewal, and ability to differentiate along lineage-specific pathways | Up to 12 months
  Descriptive statistics, such as the mean, median and range, will be used to summarize the marker across patients. The Wilcoxon signed-rank and rank sum tests will be used.
Inhibition of Notch signaling, by assessing downstream target activation | Up to 12 months
  Descriptive statistics, such as the mean, median and range, will be used to summarize the marker across patients. The Wilcoxon signed-rank and rank sum tests will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Forsyth, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (1):
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada